CLINICAL TRIAL: NCT00720941
Title: Study VEG108844, A Study of Pazopanib Versus Sunitinib in the Treatment of Subjects With Locally Advanced and/or Metastatic Renal Cell Carcinoma
Brief Title: Pazopanib Versus Sunitinib in the Treatment of Locally Advanced and/or Metastatic Renal Cell Carcinoma
Acronym: COMPARZ
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 108844; 2008-002102-19 (EudraCT Number); CPZP034A2301 (Other: Novartis); VEG108844 (Other: GlaxoSmithKline)
Record Dates: First submitted 2008-07-22; First posted 2008-07-23 (Estimated); Results first posted 2013-06-17 (Estimated); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Carcinoma, Renal Cell
Keywords: SUTENT; Locally advanced and/or metastatic renal cell carcinoma; Pazopanib; Sunitinib; GW786034; Renal cell carcinoma
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — pazopanib; Sunitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Sunitinib (Active Comparator): Control arm
  Interventions: Drug: Sunitinib
- Pazopanib (Experimental): Experimental arm
  Interventions: Drug: Pazopanib

INTERVENTIONS:
Drug: Pazopanib — 800 mg administered once daily orally continuous dosing
  Other Names: GW786034
  Arms: Pazopanib
Drug: Sunitinib — 50 mg sunitinib to be administered in 6-week cycles: 50mg orally daily for 4 weeks followed by 2 weeks off treatment
  Arms: Sunitinib

SUMMARY:
This was a randomized, open-label, parallel group Phase III non inferiority study to evaluate the efficacy and safety of pazopanib compared with sunitinib in subjects with advanced renal cell carcinoma (RCC) who had not received prior systemic therapy for advanced or metastatic RCC.

DETAILED DESCRIPTION:
Approximately 876 eligible subjects (approximately 438 per treatment arm) were planned to be enrolled over the course of the study. However, due to higher than expected withdrawal rates and discordance rates between independent review committee (IRC) and investigator assessments of progression, the protocol was amended (Protocol Amendment 4) to increase the number of subjects to approximately 1100 total by including all subjects enrolled in CPZP034A2301 (hereafter referred as Study A2301) and CPZP034A2201 (a sub study of CPZP034A2301, hereafter referred as Study A2201 with NCT01147822).

The subjects were centrally randomized in 1:1 ratio to receive either 800mg pazopanib to be administered once daily orally continuous dosing or 50mg sunitinib to be administered in 6-week cycles: 50mg orally daily for 4 weeks followed by 2 weeks off treatment. Subjects were permitted to receive supportive care throughout the study including transfusion of blood and blood products, treatment with antibiotics, anti-emetics, anti-diarrheal agents, analgesics, erythropoietin, or bisphosphonates, when appropriate. The study treatment continued until subjects experience disease progression, unacceptable toxicity, withdraw consent, or death.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Diagnosis of renal cell carcinoma with clear-cell component histology.
* Received no prior systemic therapy (interleukin-2, interferon-alpha, chemotherapy, bevacizumab, mTOR inhibitor, sunitinib, sorafenib or other VEGF TKI) for advanced or metastatic RCC
* Locally advanced or metastatic renal cell carcinoma
* Measurable disease by CT or MRI
* Karnofsky performance scale status of >=70
* Age >=18 years
* A female is eligible to enter and participate in this study if she is of: non-childbearing or agrees to use adequate contraception.
* Adequate organ system function
* Total serum calcium concentration <12.0mg/dL
* Left ventricular ejection fraction >= lower limit of institutional normal.

Exclusion Criteria:

* Pregnant or lactating female (unless agrees to refrain from nursing throughout the treatment period and for 14 days following the last dose of study)
* History of another malignancy (unless have been disease-free for 3 years)
* History or clinical evidence of central nervous system (CNS) metastases (unless have previously-treated CNS metastases and meet all 3 of the following criteria are: are asymptomatic, have had no evidence of active CNS metastases for >=6 months prior to enrolment, and have no requirement for steroids or enzyme-inducing anticonvulsants)
* Clinically significant gastrointestinal abnormalities including, but not limited to: malabsorption syndrome, major resection of the stomach or small bowel that could affect the absorption of study drug, active peptic ulcer disease, known intraluminal metastatic lesion/s with suspected bleeding, Inflammatory bowel disease, ulcerative colitis, or other gastrointestinal conditions with increased risk of perforation, history of abdominal fistula, gastrointestinal perforation, or intra abdominal abscess within 28 days prior to beginning study treatment.
* Presence of uncontrolled infection.
* Prolongation of corrected QT interval (QTc) > 480 milliseconds
* History of any one or more of the following cardiovascular conditions within the past 12 months: cardiac angioplasty or stenting, myocardial infarction, unstable angina, coronary artery by-pass graft surgery, symptomatic peripheral vascular disease, Class III or IV congestive heart failure, as defined by the New York Heart Association
* History of cerebrovascular accident including transient ischemic attack within the past 12 months
* History of pulmonary embolism or untreated deep venous thrombosis (DVT) within the past 6 months (unless had recent DVT and have been treated with therapeutic anti-coagulating agents for at least 6 weeks)
* Poorly controlled hypertension (defined as systolic blood pressure of >=150mmHg or diastolic blood pressure of >=90mmHg). Initiation or adjustment of antihypertensive medication(s) is permitted prior to study entry
* Prior major surgery or trauma within 28 days prior to first dose of study drug and/or presence of any non-healing wound, fracture, or ulcer.
* Evidence of active bleeding or bleeding susceptibility
* Spitting/coughing up blood within 6 weeks of first dose of study drug
* Known endobronchial lesions and/or lesions infiltrating major pulmonary vessels
* Any serious and/or unstable pre-existing medical, psychiatric, or other conditions that could interfere with patient's safety, obtaining informed consent or compliance to the study.
* Use any prohibited medications within 14 days of the first dose of study medication.
* Use of an investigational agent, including an investigational anti-cancer agent, within 28 days or 5 half-lives, whichever is longer, prior to the first dose of study drug.
* Prior use of an investigational or licensed drug that targets VEGF or VEGF receptors (eg. bevacizumab, sunitinib, sorafenib, etc), or are mTOR inhibitors (eg. temsirolimus, everolimus, etc).
* Is now undergoing and/or has undergone in the 14 days immediately prior to first dose of study drug, any cancer therapy (surgery, tumor embolization, chemotherapy, radiation therapy, immunotherapy, biological therapy, or hormonal therapy)
* Any ongoing toxicity from prior anti-cancer therapy that is >Grade 1 and/or that is progressing in severity.
* Known immediate or delayed hypersensitivity reaction or idiosyncrasy to drugs chemically related to pazopanib or sunitinib.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1110 (Actual)
Dates: Start 2008-08-14 (Actual); Primary Completion 2012-05-21 (Actual); Study Completion 2021-03-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (190):
- United States (85):
  - Novartis Investigative Site, Huntsville, Alabama
  - Novartis Investigative Site, Tucson, Arizona
  - Novartis Investigative Site, Little Rock, Arkansas
  - Novartis Investigative Site, Beverly Hills, California
  - Novartis Investigative Site, Escondido, California
  - Novartis Investigative Site, Fresno, California
  - Novartis Investigative Site, Greenbrae, California
  - Novartis Investigative Site, Hayward, California
  - Novartis Investigative Site, La Jolla, California
  - Novartis Investigative Site, Los Angeles, California
  - Novartis Investigative Site, Montebello, California
  - Novartis Investigative Site, Oakland, California
  - Novartis Investigative Site, Orange, California
  - Novartis Investigative Site, Roseville, California
  - Novartis Investigative Site, Sacramento, California
  - Novartis Investigative Site, San Bernardino, California
  - Novartis Investigative Site, San Francisco, California
  - Novartis Investigative Site, San Jose, California
  - Novartis Investigative Site, Santa Clara, California
  - Novartis Investigative Site, South San Francisco, California
  - Novartis Investigative Site, Vallejo, California
  - Novartis Investigative Site, Walnut Creek, California
  - Novartis Investigative Site, Denver, Colorado
  - Novartis Investigative Site, Southington, Connecticut
  - Novartis Investigative Site, Trumbull, Connecticut
  - Novartis Investigative Site, Washington D.C., District of Columbia
  - Novartis Investigative Site, Fort Myers, Florida
  - Novartis Investigative Site, Miami, Florida
  - Novartis Investigative Site, Orlando, Florida
  - Novartis Investigative Site, Atlanta, Georgia
  - Novartis Investigative Site, Chicago, Illinois
  - Novartis Investigative Site, Elk Grove Village, Illinois
  - Novartis Investigative Site, Maywood, Illinois
  - Novartis Investigative Site, Peoria, Illinois
  - Novartis Investigative Site, Carmel, Indiana
  - Novartis Investigative Site, Indianapolis, Indiana
  - Novartis Investigative Site, Cedar Rapids, Iowa
  - Novartis Investigative Site, Louisville, Kentucky
  - Novartis Investigative Site, Paducah, Kentucky
  - Novartis Investigative Site, Annapolis, Maryland
  - Novartis Investigative Site, Boston, Massachusetts
  - Novartis Investigative Site, Worcester, Massachusetts
  - Novartis Investigative Site, Detroit, Michigan
  - Novartis Investigative Site, Duluth, Minnesota
  - Novartis Investigative Site, Minneapolis, Minnesota
  - Novartis Investigative Site, Tupelo, Mississippi
  - Novartis Investigative Site, Kansas City, Missouri
  - Novartis Investigative Site, Lincoln, Nebraska
  - Novartis Investigative Site, Las Vegas, Nevada
  - Novartis Investigative Site, Lebanon, New Hampshire
  - Novartis Investigative Site, Hackensack, New Jersey
  - Novartis Investigative Site, Buffalo, New York
  - Novartis Investigative Site, New York, New York
  - Novartis Investigative Site, Hickory, North Carolina
  - Novartis Investigative Site, Raleigh, North Carolina
  - Novartis Investigative Site, Cincinnati, Ohio
  - Novartis Investigative Site, Cleveland, Ohio
  - Novartis Investigative Site, Columbus, Ohio
  - Novartis Investigative Site, Dayton, Ohio
  - Novartis Investigative Site, Oklahoma City, Oklahoma
  - Novartis Investigative Site, Tulsa, Oklahoma
  - Novartis Investigative Site, Eugene, Oregon
  - Novartis Investigative Site, Portland, Oregon
  - Novartis Investigative Site, Philadelphia, Pennsylvania
  - Novartis Investigative Site, Charleston, South Carolina
  - Novartis Investigative Site, Greenville, South Carolina
  - Novartis Investigative Site, Mt. Pleasant, South Carolina
  - Novartis Investigative Site, Chattanooga, Tennessee
  - Novartis Investigative Site, Nashville, Tennessee
  - Novartis Investigative Site, Arlington, Texas
  - Novartis Investigative Site, Bedford, Texas
  - Novartis Investigative Site, Corpus Christi, Texas
  - Novartis Investigative Site, Dallas, Texas
  - Novartis Investigative Site, Fort Worth, Texas
  - Novartis Investigative Site, Lubbock, Texas
  - Novartis Investigative Site, Round Rock, Texas
  - Novartis Investigative Site, San Antonio, Texas
  - Novartis Investigative Site, Tyler, Texas
  - Novartis Investigative Site, Webster, Texas
  - Novartis Investigative Site, Wichita Falls, Texas
  - Novartis Investigative Site, Charlottesville, Virginia
  - Novartis Investigative Site, Hampton, Virginia
  - Novartis Investigative Site, Richmond, Virginia
  - Novartis Investigative Site, Salem, Virginia
  - Novartis Investigative Site, Seattle, Washington
- Australia (9):
  - Novartis Investigative Site, Camperdown, New South Wales
  - Novartis Investigative Site, Kogarah, New South Wales
  - Novartis Investigative Site, Randwick, New South Wales
  - Novartis Investigative Site, Waratah, New South Wales
  - Novartis Investigative Site, Westmead, New South Wales
  - Novartis Investigative Site, Bedford Park, South Australia
  - Novartis Investigative Site, Hobart, Tasmania
  - Novartis Investigative Site, Heidelberg, Victoria
  - Novartis Investigative Site, Wodonga, Victoria
- Canada (11):
  - Novartis Investigative Site, Calgary, Alberta
  - Novartis Investigative Site, Edmonton, Alberta
  - Novartis Investigative Site, Vancouver, British Columbia
  - Novartis Investigative Site, Winnipeg, Manitoba
  - Novartis Investigative Site, Moncton, New Brunswick
  - Novartis Investigative Site, Hamilton, Ontario
  - Novartis Investigative Site, London, Ontario
  - Novartis Investigative Site, Oshawa, Ontario
  - Novartis Investigative Site, Ottawa, Ontario
  - Novartis Investigative Site, Toronto, Ontario
  - Novartis Investigative Site, Montreal, Quebec
- China (5):
  - Novartis Investigative Site, Guangzhou, Guangdong
  - Novartis Investigative Site, Nanjing, Jiangsu
  - Novartis Investigative Site, Beijing
  - Novartis Investigative Site, Shanghai
  - Novartis Investigative Site, Tianjin
- Germany (21):
  - Novartis Investigative Site, Kirchheim, Baden-Wurttemberg
  - Novartis Investigative Site, Sigmaringen, Baden-Wurttemberg
  - Novartis Investigative Site, Stuttgart, Baden-Wurttemberg
  - Novartis Investigative Site, Munich, Bavaria
  - Novartis Investigative Site, Planegg, Bavaria
  - Novartis Investigative Site, Marburg, Hesse
  - Novartis Investigative Site, Offenbach, Hesse
  - Novartis Investigative Site, Hanover, Lower Saxony
  - Novartis Investigative Site, Aachen, North Rhine-Westphalia
  - Novartis Investigative Site, Bonn, North Rhine-Westphalia
  - Novartis Investigative Site, Dortmund, North Rhine-Westphalia
  - Novartis Investigative Site, Duisburg, North Rhine-Westphalia
  - Novartis Investigative Site, Düsseldorf, North Rhine-Westphalia
  - Novartis Investigative Site, Essen, North Rhine-Westphalia
  - Novartis Investigative Site, Homburg, Saarland
  - Novartis Investigative Site, Dresden, Saxony
  - Novartis Investigative Site, Leipzig, Saxony
  - Novartis Investigative Site, Plauen, Saxony
  - Novartis Investigative Site, Eisleben Lutherstadt, Saxony-Anhalt
  - Novartis Investigative Site, Magdeburg, Saxony-Anhalt
  - Novartis Investigative Site, Berlin
- Ireland (3):
  - Novartis Investigative Site, Dublin
  - Novartis Investigative Site, Galway
  - Novartis Investigative Site, Tallaght, Dublin
- Italy (7):
  - Novartis Investigative Site, Napoli, Campania
  - Novartis Investigative Site, Meldola (FC), Emilia-Romagna
  - Novartis Investigative Site, Ravenna, Emilia-Romagna
  - Novartis Investigative Site, Pordenone, Friuli Venezia Giulia
  - Novartis Investigative Site, Rome, Lazio
  - Novartis Investigative Site, Milan, Lombardy
  - Novartis Investigative Site, Arezzo, Tuscany
- Japan (12):
  - Novartis Investigative Site, Ehime
  - Novartis Investigative Site, Fukuoka
  - Novartis Investigative Site, Hokkaido
  - Novartis Investigative Site, Ibaraki
  - Novartis Investigative Site, Kanagawa
  - Novartis Investigative Site, Kyoto
  - Novartis Investigative Site, Numakunai
  - Novartis Investigative Site, Okayama
  - Novartis Investigative Site, Osaka
  - Novartis Investigative Site, Shizuoka
  - Novartis Investigative Site, Tokyo
  - Novartis Investigative Site, Yamagata
- Netherlands (8):
  - Novartis Investigative Site, Alkmaar
  - Novartis Investigative Site, Amsterdam
  - Novartis Investigative Site, Breda
  - Novartis Investigative Site, Groningen
  - Novartis Investigative Site, Sittard-geleen
  - Novartis Investigative Site, The Hague
  - Novartis Investigative Site, Tilburg
  - Novartis Investigative Site, Utrecht
- South Korea (4):
  - Novartis Investigative Site, Daegu
  - Novartis Investigative Site, Daejeon
  - Novartis Investigative Site, Goyang-si, Gyeonggi-Do
  - Novartis Investigative Site, Seoul
- Spain (6):
  - Novartis Investigative Site, Badalona
  - Novartis Investigative Site, Barakaldo (Vizcaya)
  - Novartis Investigative Site, Barcelona
  - Novartis Investigative Site, Girona
  - Novartis Investigative Site, Madrid
  - Novartis Investigative Site, Pamplona
- Sweden (3):
  - Novartis Investigative Site, Lund
  - Novartis Investigative Site, Stockholm
  - Novartis Investigative Site, Uppsala
- Taiwan (4):
  - Novartis Investigative Site, Kaohsiung Hsien
  - Novartis Investigative Site, Taichung
  - Novartis Investigative Site, Taipei
  - Novartis Investigative Site, Taoyuan District
- United Kingdom (12):
  - Novartis Investigative Site, Bristol, Gloucestershire
  - Novartis Investigative Site, Northwood, Middlesex
  - Novartis Investigative Site, Bebington, Wirral
  - Novartis Investigative Site, Birmingham
  - Novartis Investigative Site, Cambridge
  - Novartis Investigative Site, Glasgow
  - Novartis Investigative Site, Leeds
  - Novartis Investigative Site, London
  - Novartis Investigative Site, Manchester
  - Novartis Investigative Site, Nottingham
  - Novartis Investigative Site, Sheffield
  - Novartis Investigative Site, Swansea

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

REFERENCES:
- [Derived] Aldin A, Besiroglu B, Adams A, Monsef I, Piechotta V, Tomlinson E, Hornbach C, Dressen N, Goldkuhle M, Maisch P, Dahm P, Heidenreich A, Skoetz N. First-line therapy for adults with advanced renal cell carcinoma: a systematic review and network meta-analysis. Cochrane Database Syst Rev. 2023 May 4;5(5):CD013798. doi: 10.1002/14651858.CD013798.pub2. PMID 37146227
- [Derived] Sheng X, Jin J, He Z, Huang Y, Zhou A, Wang J, Ren X, Ye D, Zhang X, Qin S, Zhou F, Wang B, Guo J. Pazopanib versus sunitinib in Chinese patients with locally advanced or metastatic renal cell carcinoma: pooled subgroup analysis from the randomized, COMPARZ studies. BMC Cancer. 2020 Mar 14;20(1):219. doi: 10.1186/s12885-020-6708-8. PMID 32171288
- [Derived] Sternberg CN, Motzer RJ, Hutson TE, Choueiri TK, Kollmannsberger C, Bjarnason GA, Paul Nathan, Porta C, Grunwald V, Dezzani L, Han J, Tannir NM. COMPARZ Post Hoc Analysis: Characterizing Pazopanib Responders With Advanced Renal Cell Carcinoma. Clin Genitourin Cancer. 2019 Dec;17(6):425-435.e4. doi: 10.1016/j.clgc.2019.01.015. Epub 2019 Feb 6. PMID 31601514
- [Derived] Guo J, Jin J, Oya M, Uemura H, Takahashi S, Tatsugami K, Rha SY, Lee JL, Chung J, Lim HY, Wu HC, Chang YH, Azad A, Davis ID, Carrasco-Alfonso MJ, Nanua B, Han J, Ahmad Q, Motzer R. Safety of pazopanib and sunitinib in treatment-naive patients with metastatic renal cell carcinoma: Asian versus non-Asian subgroup analysis of the COMPARZ trial. J Hematol Oncol. 2018 May 22;11(1):69. doi: 10.1186/s13045-018-0617-1. PMID 29788981
- [Derived] Grunwald V, Dietrich M, Pond GR. Early tumor shrinkage is independently associated with improved overall survival among patients with metastatic renal cell carcinoma: a validation study using the COMPARZ cohort. World J Urol. 2018 Sep;36(9):1423-1429. doi: 10.1007/s00345-018-2297-4. Epub 2018 Apr 13. PMID 29654533
- [Derived] Beaumont JL, Salsman JM, Diaz J, Deen KC, McCann L, Powles T, Hackshaw MD, Motzer RJ, Cella D. Quality-adjusted time without symptoms or toxicity analysis of pazopanib versus sunitinib in patients with renal cell carcinoma. Cancer. 2016 Apr 1;122(7):1108-15. doi: 10.1002/cncr.29888. Epub 2016 Jan 27. PMID 27000445
- [Derived] Goldstein D, Rosenberg JE, Figlin RA, Townsend RR, McCann L, Carpenter C, Pandite L. Is change in blood pressure a biomarker of pazopanib and sunitinib efficacy in advanced/metastatic renal cell carcinoma? Eur J Cancer. 2016 Jan;53:96-104. doi: 10.1016/j.ejca.2015.10.006. Epub 2015 Dec 15. PMID 26702763
- [Derived] Sorich MJ, Kichenadasse G, Rowland A, Woodman RJ, Mangoni AA. Angiotensin system inhibitors and survival in patients with metastatic renal cell carcinoma treated with VEGF-targeted therapy: A pooled secondary analysis of clinical trials. Int J Cancer. 2016 May 1;138(9):2293-9. doi: 10.1002/ijc.29972. Epub 2016 Jan 6. PMID 26685869
- [Derived] Lai JS, Beaumont JL, Diaz J, Khan S, Cella D. Validation of a short questionnaire to measure symptoms and functional limitations associated with hand-foot syndrome and mucositis in patients with metastatic renal cell carcinoma. Cancer. 2016 Jan 15;122(2):287-95. doi: 10.1002/cncr.29655. Epub 2015 Oct 12. PMID 26457466
- [Derived] Motzer RJ, Hutson TE, Cella D, Reeves J, Hawkins R, Guo J, Nathan P, Staehler M, de Souza P, Merchan JR, Boleti E, Fife K, Jin J, Jones R, Uemura H, De Giorgi U, Harmenberg U, Wang J, Sternberg CN, Deen K, McCann L, Hackshaw MD, Crescenzo R, Pandite LN, Choueiri TK. Pazopanib versus sunitinib in metastatic renal-cell carcinoma. N Engl J Med. 2013 Aug 22;369(8):722-31. doi: 10.1056/NEJMoa1303989. PMID 23964934

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants were stratified based on Karnofsky Performance Scale scores (70 or 80; 90 or 100), Baseline levels of lactate dehydrogenase (>1.5 versus <=1.5 times the upper limit of normal [ULN]), and previous nephrectomy (yes versus no) and were randomized in a 1:1 ratio to receive either pazopanib or sunitinib.
Groups:
- Pazopanib 800 mg: Participants were administered pazopanib 800 milligrams (mg) (2 x 400 mg tablets) orally once daily (OD) continuously. Pazopanib was to be taken at least one hour before or at least two hours after a meal. Participants received study treatment until disease progression, death, unacceptable toxicity, or withdrawal of consent for any other reasons.
- Sunitinib 50 mg: Participants were administered sunitinib 50 mg orally once daily in 6-week cycles (4 weeks of treatment, followed by 2 weeks without treatment). Participants received study treatment until disease progression, death, unacceptable toxicity, or withdrawal of consent for any other reasons.
Period: Overall Study
Arm/Group | Pazopanib 800 mg | Sunitinib 50 mg
Started (All randomized subjects from Study A2301 and Study A2201 were included in the Intent-to-Treat (ITT) Population) | 557 | 553
Safety Population (All randomized subjects from Study A2301 and Study A2201 who received at least one dose of study treatment were included in the Safety Population) | 554 | 548
Completed | 485 | 481
Not Completed | 72 | 72
Not completed — Protocol Violation | 1 | 2
Not completed — Transitioned to another mechanism of continuing pazopanib or sunitinib therapy after 30SEP2013 | 8 | 7
Not completed — Lost to Follow-up | 20 | 15
Not completed — Physician Decision | 14 | 12
Not completed — Withdrawal by Subject | 29 | 36

BASELINE CHARACTERISTICS:
Groups:
- Pazopanib 800 mg: Participants were administered pazopanib 800 mg (2 x 400 mg tablets) orally OD continuously. Pazopanib was to be taken at least one hour before or at least two hours after a meal. Participants received study treatment until disease progression, death, unacceptable toxicity, or withdrawal of consent for any other reasons.
- Total: Total of all reporting groups
Arm/Group | Pazopanib 800 mg | Sunitinib 50 mg | Total
Number analyzed (Participants) | 557 | 553 | 1110
Age, Continuous [Mean (Standard Deviation); unit: Years] | 60.9 (10.89) | 61.2 (10.98) | 61.1 (10.93)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 159 | 138 | 297
  Male | 398 | 415 | 813
Race/Ethnicity, Customized [Number; unit: Participants]
  White | 349 | 358 | 707
  Asian | 194 | 188 | 382
  African American/African Heritage | 10 | 5 | 15
  American Indian or Alaska Native | 3 | 0 | 3
  American Indian or Alaska Native & White | 0 | 1 | 1
  Unknown | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival (PFS)
Description: PFS was defined as the interval between the date of randomization and the earliest date of progressive disease (PD), as defined by the Independent Review Committee (IRC), or death due to any cause. The IRC defined PD per Response Evaluation Criteria in Solid Tumors (RECIST), Version 1. Per RECIST, PD is defined as a >=20% increase in the sum of the longest diameter of target lesions, taking as reference the smallest sum longest diameter recorded since the treatment started or the appearance of >=1 new lesion.
Time Frame: From randomization until the earliest date of disease progression or date of death from any cause, assessed up to approximately 39 months
Population: Intent-to-Treat (ITT) Population. Analysis was based on the assigned randomized treatment, not on the actual treatment received/not received. Participants who had neither progressed nor died were censored at the date of the last adequate tumor assessment at the time of the cut-off.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pazopanib 800 mg | Sunitinib 50 mg
Number analyzed (Participants) | 557 | 553
Months | 8.4 [8.3 to 10.9] | 9.5 [8.3 to 11.1]
Statistical Analysis 1: Comparison: Pazopanib 800 mg vs Sunitinib 50 mg; Test type: Non-Inferiority or Equivalence — Non-inferiority is defined as excluding a difference of greater than 25% in the hazards. The upper limit of the 95% confidence interval must be <1.25; Hazard Ratio (HR) = 1.0466, 95% CI 2-sided [0.8982 to 1.2195] — The HR is estimated by the Cox regression model using treatment stratification factors as covariates. The HR is adjusted for Karnofsky Performance Scale scores, prior nephrectomy, and Baseline levels of lactate dehydrogenase (<=1.5xULN, >1.5xULN)

2. Secondary Outcome: Overall Survival
Description: Overall survival was defined as the time from randomization until death due to any cause.
Time Frame: From randomization until date of death from any cause, assessed up to approximately 62 months
Population: Intent-to-Treat (ITT) Population. Analysis was based on the assigned randomized treatment, not on the actual treatment received/not received. Participants who had not died were censored at the date of the last adequate tumor assessment at the time of the cut-off.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pazopanib 800 mg | Sunitinib 50 mg
Number analyzed (Participants) | 557 | 553
Months | 28.3 [26.0 to 35.5] | 29.1 [25.4 to 33.1]

3. Secondary Outcome: Overall Response Rate (ORR) as Assessed by Independent Review
Description: The number of participants with evidence of Complete Response (CR) (the disappearance of all target and non-target lesions), Partial Response (PR) (at least a 30% decrease in the sum of the longest diameters [LD] of target lesions, taking as a reference the Baseline sum LD), Stable Disease (small changes that do not meet previously given criteria, taking as reference the smallest sum LD since the treatment started), or Progressive Disease (a >=20% increase in the sum of the LD of target lesions, taking as a reference the smallest sum LD recorded since the treatment started) was evaluated by an independent review per RECIST, Version 1.
Time Frame: From randomization until date of radiographic progression or date of death from any cause, whichever comes first, assessed up to approximately 39 months
Population: Intent-to-Treat (ITT) Population. Analysis was based on the assigned randomized treatment, not on the actual treatment received/not received.
Measure: Count of Participants; unit: Participants
Arm/Group | Pazopanib 800 mg | Sunitinib 50 mg
Number analyzed (Participants) | 557 | 553
Participants
  Complete Response | 1 | 3
  Partial Response | 170 | 134
  Stable Disease | 216 | 242
  Progressive Disease | 97 | 105
  Unknown | 73 | 69

4. Secondary Outcome: Time to Response
Description: Time to response was defined as the time from the start of treatment until the first documented evidence of CR (the disappearance of all target and non-target lesions) or PR (at least a 30% decrease in the sum of the LD of target lesions, taking as a reference the Baseline sum LD), whichever comes first. CR and PR were evaluated by an independent review per RECIST, Version 1.
Time Frame: as for outcome 3
Population: Intent-to-Treat (ITT) Population. Analysis was based on the assigned randomized treatment, not on the actual treatment received/not received. Only those participants who experienced either a confirmed CR or a PR were analyzed.
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | Pazopanib 800 mg | Sunitinib 50 mg
Number analyzed (Participants) | 171 | 137
Weeks | 11.9 [11.3 to 12.1] | 17.4 [12.7 to 18.0]

5. Secondary Outcome: Duration of Response (DOR)
Description: DOR was defined as the time from the first documented evidence of response (CR or PR) until the first documented sign of disease progression (a >=20% increase in the sum of the longest diameter of target lesions, taking as reference the smallest sum longest diameter recorded since the treatment started or the appearance of >=1 new lesion) or death, if sooner. CR=the disappearance of all target and non-target lesions. PR=at least a 30% decrease in the sum of the LD of target lesions, taking as a reference the Baseline sum LD.
Time Frame: From the date of the first documented response (CR or PR) to the date of first documented progression or death due to any cause, assessed up to approximately 39 months
Population: Intent-to-Treat (ITT) Population. Analysis was based on the assigned randomized treatment, not on the actual treatment received/not received. Only those participants who had either a confirmed CR or PR were analyzed.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pazopanib 800 mg | Sunitinib 50 mg
Number analyzed (Participants) | 171 | 137
Months | 13.8 [12.2 to 16.4] | 18.0 [14.3 to 22.1]

6. Secondary Outcome: Number of Participants With Adverse Events
Description: The distribution of adverse events was done via the analysis of frequencies for Adverse Event (AEs) and Serious Adverse Event (SAEs), through the monitoring of relevant clinical and laboratory safety parameters.
Time Frame: From study treatment start date till 28 days safety follow-up, assessed up to approximately 152 months
Population: Safety Population: all randomized participants who received at least one dose of study medication, according to the actual treatment received.
Measure: Count of Participants; unit: Participants
Arm/Group | Pazopanib 800 mg | Sunitinib 50 mg
Number analyzed (Participants) | 554 | 548
Participants
  Adverse Events (AEs) | 551 | 535
  Serious Adverse Events (SAEs) | 242 | 227

7. Secondary Outcome: Change From Baseline in Functional Assessment of Chronic Illness Therapy-Fatigue (FACIT-F) Scale Scores at Day 28 of Cycles 1-4
Description: FACIT Fatigue Subscale is a short, 13-item, easy to administer tool that measures an individual's level of fatigue during their usual daily activities over the past week. The level of fatigue is measured on a four point Likert scale (4 = not at all fatigued to 0 = very much fatigued). The total score range is from 0-52. The higher the score, the lower the fatigue level.
Time Frame: Baseline (predose), Day 28 of Cycles 1-4 (average of Weeks 4, 10, 16, and 22, respectively)
Population: Intent-to-Treat (ITT) Population. Analysis was based on the assigned randomized treatment, not on the actual treatment received/not received. Some participants were missing scores at Baseline and were excluded from the analysis. Participants missing scores at some of the other early time points were excluded from the analysis at those time points.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Pazopanib 800 mg | Sunitinib 50 mg
Number analyzed (Participants) | 353 | 375
Scores on a scale
  Week 4 (n=353,375) | -5.3 (11.00) | -6.7 (10.93)
  Week 10 (n=293,330): number analyzed (Participants) | 293 | 330
  Week 10 (n=293,330) | -4.0 (10.28) | -6.3 (10.65)
  Week 16 (n=273,280): number analyzed (Participants) | 273 | 280
  Week 16 (n=273,280) | -3.8 (10.13) | -6.9 (11.16)
  Week 22 (n=227,240): number analyzed (Participants) | 227 | 240
  Week 22 (n=227,240) | -2.9 (9.77) | -6.5 (10.51)

8. Secondary Outcome: Change From Baseline in the FACT-Kidney Symptom Index-19 (FKSI-19) Scale Disease-related Symptoms-physical (DRS-P) Domain Score at Day 28 of Cycles 1-4
Description: Health outcome and quality of life as measured by NCCN/FACT FKSI-19 questionnaire. The FKSI-19 is a disease-specific instrument that measures disease and treatment-related symptoms specifically in renal cancer patients in 4 domains (Disease-Related Symptoms - Physical (FKSI-DRS-P), Disease-Related Symptoms - Emotional (FKSI-DRS-E), Treatment Side-Effects (FKSI-TSE), Function/Well-Being (FKSI-FWB)) experienced in the past 7 days. Participants are asked to respond to a total of 19 questions regarding symptoms, side effects, and well being by using a 5-point scale (0=not at all, 1=a little bit, 2=somewhat, 3=quite a bit, 4=very much; possible total score of 0 to 76). A negative mean indicates a worsening of condition.
Time Frame: Baseline (predose), Day 28 of Cycles 1-4 (average of Weeks 4, 10, 16, and 22, respectively)
Population: Intent-to-Treat (ITT) Population. Analysis was based on the assigned randomized treatment, not on the actual treatment received/not received. Some participants were missing scores at Baseline and were excluded from the analysis. Participants missing scores at other early time points were excluded from the analysis at those time points. Change from Baseline was calculated as the assessment week value minus the Baseline value.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Pazopanib 800 mg | Sunitinib 50 mg
Number analyzed (Participants) | 358 | 378
Scores on a scale
  Week 4 (n=358,378) | -2.9 (6.39) | -3.9 (6.87)
  Week 10 (n=296,336): number analyzed (Participants) | 296 | 336
  Week 10 (n=296,336) | -2.3 (6.69) | -3.2 (6.76)
  Week 16 (n=269,283): number analyzed (Participants) | 269 | 283
  Week 16 (n=269,283) | -2.6 (6.70) | -3.2 (6.61)
  Week 22 (n=224,238): number analyzed (Participants) | 224 | 238
  Week 22 (n=224,238) | -1.3 (6.29) | -2.7 (6.42)

9. Secondary Outcome: Change From Baseline in the FACT-Kidney Symptom Index-19 (FKSI-19) Scale Disease Related Symptoms-emotional (DRS-E) Domain Score at Day 28 of Cycles 1-4
Description: as for outcome 8
Time Frame: Baseline (predose), Day 28 of Cycles 1-4 (average of Weeks 4, 10, 16, and 22, respectively)
Population: Intent-to-Treat (ITT) Population. Analysis was based on the assigned randomized treatment, not on the actual treatment received/not received. Some participants were missing scores at Baseline and were excluded from the analysis. Participants missing scores at other early time points were excluded from the analysis at those time points.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Pazopanib 800 mg | Sunitinib 50 mg
Number analyzed (Participants) | 344 | 367
Scores on a scale
  Week 4 (n=344,367) | 0.3 (1.31) | 0.4 (1.22)
  Week 10 (n=287,329): number analyzed (Participants) | 287 | 329
  Week 10 (n=287,329) | 0.4 (1.33) | 0.5 (1.32)
  Week 16 (n=260,277): number analyzed (Participants) | 260 | 277
  Week 16 (n=260,277) | 0.5 (1.39) | 0.6 (1.30)
  Week 22 (n=220,233): number analyzed (Participants) | 220 | 233
  Week 22 (n=220,233) | 0.6 (1.27) | 0.6 (1.20)

10. Secondary Outcome: Change From Baseline in the FACT-Kidney Symptom Index-19 (FKSI-19) Scale Treatment Side Effects (TSE) Domain Score at Day 28 of Cycles 1-4
Description: as for outcome 8
Time Frame: Baseline (predose), Day 28 of Cycles 1-4 (average of Weeks 4, 10, 16, and 22, respectively)
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Pazopanib 800 mg | Sunitinib 50 mg
Number analyzed (Participants) | 326 | 350
Scores on a scale
  Week 4 (n=326,350) | -1.5 (2.45) | -2.0 (2.35)
  Week 10 (n=267,305): number analyzed (Participants) | 267 | 305
  Week 10 (n=267,305) | -1.9 (2.66) | -2.4 (2.62)
  Week 16 (n=244,254): number analyzed (Participants) | 244 | 254
  Week 16 (n=244,254) | -2.1 (2.79) | -2.8 (2.46)
  Week 22 (n=201,218): number analyzed (Participants) | 201 | 218
  Week 22 (n=201,218) | -2.4 (2.75) | -2.4 (2.33)

11. Secondary Outcome: Change From Baseline in the FACT-Kidney Symptom Index-19 (FKSI-19) Scale Functional Well Being (FWB) Domain Score at Day 28 of Cycles 1-4
Description: as for outcome 8
Time Frame: Baseline (predose), Day 28 of Cycles 1-4 (average of Weeks 4, 10, 16, and 22, respectively)
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Pazopanib 800 mg | Sunitinib 50 mg
Number analyzed (Participants) | 357 | 378
Scores on a scale
  Week 4 (n=357,378) | -1.0 (4.01) | -1.3 (3.63)
  Week 10 (n=298,331): number analyzed (Participants) | 298 | 331
  Week 10 (n=298,331) | -0.6 (4.00) | -1.1 (3.94)
  Week 16 (n=267,278): number analyzed (Participants) | 267 | 278
  Week 16 (n=267,278) | -0.8 (4.08) | -1.0 (3.96)
  Week 22 (n=228,234): number analyzed (Participants) | 228 | 234
  Week 22 (n=228,234) | -0.7 (3.93) | -1.0 (3.82)

12. Secondary Outcome: Change From Baseline in the FACT-Kidney Symptom Index-19 (FKSI-19) Scale Total Score at Day 28 of Cycles 1-4
Description: as for outcome 8
Time Frame: Baseline (predose), Day 28 of Cycles 1-4 (average of Weeks 4, 10, 16, and 22, respectively)
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Pazopanib 800 mg | Sunitinib 50 mg
Number analyzed (Participants) | 358 | 379
Scores on a scale
  Week 4 (n=358,379) | -5.0 (10.82) | -6.6 (10.55)
  Week 10 (n=296,337): number analyzed (Participants) | 296 | 337
  Week 10 (n=296,337) | -4.2 (10.95) | -6.3 (11.21)
  Week 16 (n=267,284): number analyzed (Participants) | 267 | 284
  Week 16 (n=267,284) | -4.8 (11.13) | -6.3 (10.67)
  Week 22 (n=225,238): number analyzed (Participants) | 225 | 238
  Week 22 (n=225,238) | -3.7 (10.49) | -5.5 (10.13)

13. Secondary Outcome: Change From Baseline in the Supplementary Quality of Life Questions (SQLQ) Scale Worst Soreness Scores at Day 28 of Cycles 1-4
Description: The SQLQ scale consists of 5 items that assess the worst mouth and throat, hand, and foot soreness, as well as limitations due to mouth/throat and foot soreness. Participants were asked to assess their worst mouth/throat, hand, and foot soreness by answering the question of " In the past 4 weeks, what was your worst mouth/throat, hand, and foot soreness?" by using the following 4-point scale: 0, I never had any soreness; 1, I had a little bit of soreness; 2, I had quite a lot of soreness; 3, I had severe soreness. A positive mean change from Baseline represents a worsening of condition.
Time Frame: Baseline (predose), Day 28 of Cycles 1-4 (average of Weeks 4, 10, 16, and 22, respectively)
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Pazopanib 800 mg | Sunitinib 50 mg
Number analyzed (Participants) | 202 | 184
Scores on a scale
  Mouth and Throat Soreness, Week 4 (n=202,180): number analyzed (Participants) | 202 | 180
  Mouth and Throat Soreness, Week 4 (n=202,180) | 0.4 (0.87) | 1.0 (0.99)
  Mouth and Throat Soreness, Week 10 (n=164,155): number analyzed (Participants) | 164 | 155
  Mouth and Throat Soreness, Week 10 (n=164,155) | 0.4 (0.88) | 0.9 (0.99)
  Mouth and Throat Soreness, Week 16 (n=137,138): number analyzed (Participants) | 137 | 138
  Mouth and Throat Soreness, Week 16 (n=137,138) | 0.3 (0.73) | 0.8 (0.89)
  Mouth and Throat Soreness, Week 22 (n=120,117): number analyzed (Participants) | 120 | 117
  Mouth and Throat Soreness, Week 22 (n=120,117) | 0.2 (0.75) | 0.8 (0.81)
  Hand Soreness, Week 4 (n=200,184): number analyzed (Participants) | 200 | 184
  Hand Soreness, Week 4 (n=200,184) | 0.2 (0.71) | 0.3 (0.72)
  Hand Soreness, Week 10 (n=164,153): number analyzed (Participants) | 164 | 153
  Hand Soreness, Week 10 (n=164,153) | 0.3 (0.84) | 0.7 (0.85)
  Hand Soreness, Week 16 (n=139,136): number analyzed (Participants) | 139 | 136
  Hand Soreness, Week 16 (n=139,136) | 0.4 (0.76) | 0.6 (0.80)
  Hand Soreness, Week 22 (n=123,115): number analyzed (Participants) | 123 | 115
  Hand Soreness, Week 22 (n=123,115) | 0.3 (0.69) | 0.6 (0.82)
  Foot Soreness, Week 4 (n=199,182): number analyzed (Participants) | 199 | 182
  Foot Soreness, Week 4 (n=199,182) | 0.2 (0.86) | 0.4 (0.80)
  Foot Soreness, Week 10 (n=163,153): number analyzed (Participants) | 163 | 153
  Foot Soreness, Week 10 (n=163,153) | 0.3 (1.00) | 0.6 (0.99)
  Foot Soreness, Week 16 (n=140,136): number analyzed (Participants) | 140 | 136
  Foot Soreness, Week 16 (n=140,136) | 0.3 (1.07) | 0.8 (0.99)
  Foot Soreness, Week 22 (n=123,116): number analyzed (Participants) | 123 | 116
  Foot Soreness, Week 22 (n=123,116) | 0.3 (1.04) | 0.9 (0.96)

14. Secondary Outcome: Change From Baseline in the Supplementary Quality of Life Questions (SQLQ) Limitations Due to Mouth and Throat Soreness Score at Day 28 of Cycles 1-4
Description: The SQLQ consists of 5 items assessing the worst mouth/throat, hand, and foot soreness, and limitations due to mouth/throat and foot soreness. Participants assessed the limitations caused by their mouth/throat soreness by answering the question of "In the past 4 weeks, how much did your worst mouth/throat soreness limit you in the following activities: swallowing/eating/drinking/talking/sleeping" by using the following 4-point scale: 0, not limited; 1, limited a little; 2, limited a lot; 3, unable to do. The overall limitation score (15=best; 0=worst), based on the individual scores for the 5 activities, is derived as follows: the actual scores were rescored by subtracting the actual score from "3" for each of the 5 categories. A high score indicates less limitation. Change from Baseline was calculated as the assessment week value minus the Baseline value. A negative mean change from Baseline represents a worsening of condition.
Time Frame: Baseline (predose), Day 28 of Cycles 1-4 (average of Weeks 4, 10, 16, and 22, respectively)
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Pazopanib 800 mg | Sunitinib 50 mg
Number analyzed (Participants) | 177 | 170
Scores on a scale
  Week 4 (n=177,170) | -0.9 (2.09) | -1.8 (2.91)
  Week 10 (n=144,137): number analyzed (Participants) | 144 | 137
  Week 10 (n=144,137) | -0.9 (1.91) | -1.8 (3.06)
  Week 16 (n=125,122): number analyzed (Participants) | 125 | 122
  Week 16 (n=125,122) | -0.6 (1.56) | -1.3 (2.30)
  Week 22 (n=111,107): number analyzed (Participants) | 111 | 107
  Week 22 (n=111,107) | -0.4 (1.67) | -1.4 (1.85)

15. Secondary Outcome: Change From Baseline in the Supplementary Quality of Life Questions (SQLQ) Limitations Due to Foot Soreness Scores at Day 28 of Cycles 1-4
Description: The SQLQ consists of 5 items assessing the worst mouth/throat, hand, and foot soreness, and limitations due to mouth/throat and foot soreness. Participants assessed the limitations caused by their foot soreness by answering the question of "In the past 4 weeks, how much did your worst foot soreness limit you in each of the following activities: standing/walking/climbing stairs/sleeping/ability to do usual activities" by using the following 4-point scale: 0, not limited; 1, limited a little; 2, limited a lot; 3, unable to do. The overall limitation score (15=best; 0=worst), based on the individual scores for the 5 activities, is derived as follows: the actual scores were rescored by subtracting the actual score from "3" for each of the 5 categories. A high score indicates less limitation. Change from Baseline was calculated as the assessment week value minus the Baseline value. A negative mean change from Baseline represents a worsening of condition.
Time Frame: Baseline (predose), Day 28 of Cycles 1-4 (average of Weeks 4, 10, 16, and 22, respectively)
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Pazopanib 800 mg | Sunitinib 50 mg
Number analyzed (Participants) | 170 | 163
Scores on a scale
  Week 4 (n=170,163) | -0.6 (2.94) | -1.0 (2.94)
  Week 10 (n=133,136): number analyzed (Participants) | 133 | 136
  Week 10 (n=133,136) | -1.1 (3.02) | -1.5 (3.76)
  Week 16 (n=114,126): number analyzed (Participants) | 114 | 126
  Week 16 (n=114,126) | -1.2 (3.42) | -2.2 (3.50)
  Week 22 (n=105,108): number analyzed (Participants) | 105 | 108
  Week 22 (n=105,108) | -1.3 (3.25) | -2.1 (3.52)

16. Secondary Outcome: Summary of Analysis for the Cancer Treatment Satisfaction Questionnaire (CTSQ) Score at Day 28 of Cycles 1-4
Description: The CTSQ assesses 3 domains related to the participant's satisfaction with cancer therapy: Expectations of Therapy (ET), Feelings about Side Effects (FSE), and Satisfaction with Therapy (SWT). Participants shared their thoughts on their cancer therapy (9 questions), their satisfaction with their most recently administered cancer therapy (6 questions), and if they would take the same cancer therapy if given the choice to do so again. All questions were assessed on a 5-point scale; 1, never; 5, always. Scores were averaged and transformed to a 0-100 scale; higher scores represent better treatment satisfaction.
Time Frame: Day 28 of Cycles 1-4 (average of Weeks 4, 10, 16, and 22, respectively)
Population: Intent-to-Treat (ITT) Population. Analysis was based on the assigned randomized treatment, not on the actual treatment received/not received. Participants missing scores at early time points were excluded from the analysis at those time points. Mean total score was calculated at each assessment week.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Pazopanib 800 mg | Sunitinib 50 mg
Number analyzed (Participants) | 383 | 386
Scores on a scale
  ET, Week 4 (n=383,386) | 71.7 (22.13) | 71.3 (22.38)
  ET, Week 10 (n=321,346): number analyzed (Participants) | 321 | 346
  ET, Week 10 (n=321,346) | 73.4 (21.62) | 73.4 (19.37)
  ET, Week 16 (n=296,293): number analyzed (Participants) | 296 | 293
  ET, Week 16 (n=296,293) | 73.9 (21.56) | 72.9 (21.43)
  ET, Week 22 (n=250,250): number analyzed (Participants) | 250 | 250
  ET, Week 22 (n=250,250) | 73.0 (21.40) | 73.4 (20.43)
  FSE, Week 4 (n=340,360): number analyzed (Participants) | 340 | 360
  FSE, Week 4 (n=340,360) | 66.3 (24.00) | 58.5 (23.59)
  FSE, Week 10 (n=298,323): number analyzed (Participants) | 298 | 323
  FSE, Week 10 (n=298,323) | 66.0 (23.09) | 56.0 (22.23)
  FSE, Week 16 (n=274,277): number analyzed (Participants) | 274 | 277
  FSE, Week 16 (n=274,277) | 65.0 (23.01) | 56.6 (22.02)
  FSE, Week 22 (n=235, 232): number analyzed (Participants) | 235 | 232
  FSE, Week 22 (n=235, 232) | 67.1 (22.62) | 57.8 (21.28)
  SWT, Week 4 (n=355,374): number analyzed (Participants) | 355 | 374
  SWT, Week 4 (n=355,374) | 80.9 (15.49) | 79.0 (15.23)
  SWT, Week 10 (n=309,336): number analyzed (Participants) | 309 | 336
  SWT, Week 10 (n=309,336) | 84.5 (13.74) | 80.4 (15.15)
  SWT, Week 16 (n=287,284): number analyzed (Participants) | 287 | 284
  SWT, Week 16 (n=287,284) | 85.3 (14.77) | 80.5 (15.08)
  SWT, Week 22 (n=241,240): number analyzed (Participants) | 241 | 240
  SWT, Week 22 (n=241,240) | 85.4 (13.48) | 81.4 (15.04)

17. Secondary Outcome: Mean Number of Non-study Medical Visits, Telephone Consultations, Hospital Days, and Emergency Room (ER) Visits Per 30 Days Through Week 24
Description: Non-study medical visits were defined as the sum of primary care physician visits, nurse practitioner/physician's assistant/nurse visits, and medical or surgical specialist visits. Days hospitalized were defined as the sum of days in the general ward and days in intensive care. The number of telephone consultations and ER visits was assessed via individual questions on the electronic Case Report Form. The endpoint was totaled through Week 24, divided by the number of days on treatment for each participant, then multiplied by 30 days to get the number of visits per 30 days.
Time Frame: From Day 1 up to Week 24
Population: Intent-to-Treat (ITT) Population. Analysis was based on the assigned randomized treatment, not on the actual treatment received/not received. Only those participants who had non-study medical visits, telephone consultations, days in the hospital, and ER visits were analyzed.
Measure: Mean (Standard Deviation); unit: events per 30 days
Arm/Group | Pazopanib 800 mg | Sunitinib 50 mg
Number analyzed (Participants) | 429 | 432
events per 30 days
  Non-Study Medical Visits | 0.726 (1.472) | 0.779 (1.690)
  Telephone Consultations | 0.279 (0.718) | 0.312 (0.656)
  Hospital Days | 0.402 (2.273) | 0.562 (2.187)
  ER Visits | 0.037 (0.156) | 0.067 (0.195)

18. Secondary Outcome: Mean Number of Laboratory Visits, Radiology Visits, Home Healthcare Visits, and Medical Procedures at Day 28 of Cycles 1-4
Description: The number of non-study laboratory visits (NSLVs), non-study radiology visits (NSRVs), and home healthcare visits (HHVs) were each collected as a single question on the eCRF. The number of non-study medical or surgical procedures (MSPs) was defined as the sum of procedures performed at outpatient or physician clinics, as well as those performed during any inpatient hospitalization.
Time Frame: Day 28 of Cycles 1-4 (average of Weeks 4, 10, 16, and 22, respectively)
Population: Intent-to-Treat (ITT) Population. Analysis was based on the assigned randomized treatment, not on the actual treatment received/not received. Only those participants who had NSLVs, NSRVs, HHVs, and medical procedures were analyzed.
Measure: Mean (Standard Deviation); unit: visits
Arm/Group | Pazopanib 800 mg | Sunitinib 50 mg
Number analyzed (Participants) | 429 | 432
visits
  NSLV, Cycle 1 (n=417,414): number analyzed (Participants) | 417 | 414
  NSLV, Cycle 1 (n=417,414) | 0.3 (1.25) | 0.3 (1.14)
  NSLV, Cycle 2 (n=345,363): number analyzed (Participants) | 345 | 363
  NSLV, Cycle 2 (n=345,363) | 0.3 (0.97) | 0.4 (1.35)
  NSLV, Cycle 3 (n=299,304): number analyzed (Participants) | 299 | 304
  NSLV, Cycle 3 (n=299,304) | 0.2 (0.67) | 0.2 (0.58)
  NSLV, Cycle 4 (n=265,254): number analyzed (Participants) | 265 | 254
  NSLV, Cycle 4 (n=265,254) | 0.1 (0.49) | 0.1 (0.47)
  NSRV, Cycle 1 (n=419,414): number analyzed (Participants) | 419 | 414
  NSRV, Cycle 1 (n=419,414) | 0.1 (0.44) | 0.1 (0.56)
  NSRV, Cycle 2 (n=348,364): number analyzed (Participants) | 348 | 364
  NSRV, Cycle 2 (n=348,364) | 0.1 (0.36) | 0.1 (0.88)
  NSRV, Cycle 3 (n=299,305): number analyzed (Participants) | 299 | 305
  NSRV, Cycle 3 (n=299,305) | 0.0 (0.28) | 0.1 (0.33)
  NSRV, Cycle 4 (n=266,255): number analyzed (Participants) | 266 | 255
  NSRV, Cycle 4 (n=266,255) | 0.0 (0.24) | 0.1 (0.46)
  HHV, Cycle 1 (n=418,411): number analyzed (Participants) | 418 | 411
  HHV, Cycle 1 (n=418,411) | 0.0 (0.44) | 0.1 (0.77)
  HHV, Cycle 2 (n=343,363): number analyzed (Participants) | 343 | 363
  HHV, Cycle 2 (n=343,363) | 0.1 (0.52) | 0.1 (0.64)
  HHV, Cycle 3 (n=298,304): number analyzed (Participants) | 298 | 304
  HHV, Cycle 3 (n=298,304) | 0.1 (0.72) | 0.0 (0.37)
  HHV, Cycle 4 (n=265,254): number analyzed (Participants) | 265 | 254
  HHV, Cycle 4 (n=265,254) | 0.0 (0.49) | 0.1 (1.77)
  NSP, Cycle 1 (n=417,413): number analyzed (Participants) | 417 | 413
  NSP, Cycle 1 (n=417,413) | 0.2 (0.69) | 0.3 (2.52)
  NSP, Cycle 2 (n=344,363): number analyzed (Participants) | 344 | 363
  NSP, Cycle 2 (n=344,363) | 0.2 (0.68) | 0.2 (1.17)
  NSP, Cycle 3 (n=298,304): number analyzed (Participants) | 298 | 304
  NSP, Cycle 3 (n=298,304) | 0.2 (0.60) | 0.3 (1.98)
  NSP, Cycle 4 (n=266,254): number analyzed (Participants) | 266 | 254
  NSP, Cycle 4 (n=266,254) | 0.2 (0.85) | 0.3 (1.73)

19. Other Pre Specified Outcome: All Collected Deaths
Description: Pre-treatment deaths were collected from day of participant's informed consent to the day before first dose of study medication.
  On-treatment deaths were collected from first dose of study medication to 28 days after last dose of study medication (on-treatment), up to approximately 129 months.
  Deaths were collected in the post treatment survival follow up from 29 days after last dose of study medication until the end of the study, up to approximately 152 months.
Time Frame: Pre-treatment deaths: Up to 21 days prior to treatment. On-treatment deaths: Up to 129 months. Post-treatment deaths: up to 152 months.
Population: Intent-to-Treat (ITT) Population
Measure: Count of Participants; unit: Participants
Arm/Group | Pazopanib 800 mg | Sunitinib 50 mg
Number analyzed (Participants) | 557 | 553
Participants
  Pre-treatment deaths | 0 | 0
  On-treatment deaths: number analyzed (Participants) | 554 | 548
  On-treatment deaths | 25 | 22
  Post-treatment deaths: number analyzed (Participants) | 529 | 526
  Post-treatment deaths | 310 | 312
  All deaths | 335 | 334

ADVERSE EVENTS:
Time Frame: Adverse Events (AEs) were collected from first dose of study medication until the last dose plus 28 days post-treat follow-up, assessed up to approximately 129 months. Deaths were recorded from study start date until end of survival follow-up phase (end of study), assessed up to approximately 152 months.
Description: Deaths in the post-treatment survival follow-up were not considered adverse events. The total number at risk in the post-treatment survival included patients who entered this period. All-cause Mortality was assessed for all participants enrolled in the study, while Serious and Other Adverse Events were assessed for all participants who received at least one dose of the study medication.
Groups:
- Pazopanib 800 mg: Pazopanib 800 mg: Events up to 28 days post-treatment
- Sunitinib 50 mg: Sunitinib 50 mg: Events up to 28 days post-treatment
- Pazopanib 800 mg (Post-Treatment): Pazopanib 800 mg (Post-Treatment) - Deaths in the post-treatment survival follow-up were not considered adverse events.
- Sunitinib 50 mg (Post-Treatment): Sunitinib 50 mg (Post-Treatment) - Deaths in the post-treatment survival follow-up were not considered adverse events.
Arm/Group | Pazopanib 800 mg | Sunitinib 50 mg | Pazopanib 800 mg (Post-Treatment) | Sunitinib 50 mg (Post-Treatment)
All-Cause Mortality (participants affected / at risk) | 25/557 | 22/553 | 310/529 | 312/526
Serious Adverse Events (participants affected / at risk) | 242/554 | 227/548 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 541/554 | 535/548 | 0/0 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pazopanib 800 mg (N=554) | Sunitinib 50 mg (N=548) | Pazopanib 800 mg (Post-Treatment) (N=0) | Sunitinib 50 mg (Post-Treatment) (N=0)
Anaemia (Blood and lymphatic system disorders) | 9 | 9 | NA | NA
Febrile neutropenia (Blood and lymphatic system disorders) | 2 | 0 | NA | NA
Immune thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1 | NA | NA
Lymphopenia (Blood and lymphatic system disorders) | 0 | 1 | NA | NA
Microangiopathic haemolytic anaemia (Blood and lymphatic system disorders) | 0 | 1 | NA | NA
Neutropenia (Blood and lymphatic system disorders) | 2 | 7 | NA | NA
Polycythaemia (Blood and lymphatic system disorders) | 2 | 0 | NA | NA
Thrombocytopenia (Blood and lymphatic system disorders) | 4 | 24 | NA | NA
Acute myocardial infarction (Cardiac disorders) | 3 | 2 | NA | NA
Angina pectoris (Cardiac disorders) | 2 | 0 | NA | NA
Angina unstable (Cardiac disorders) | 1 | 1 | NA | NA
Atrial fibrillation (Cardiac disorders) | 1 | 0 | NA | NA
Atrial thrombosis (Cardiac disorders) | 0 | 1 | NA | NA
Bradycardia (Cardiac disorders) | 0 | 1 | NA | NA
Cardiac failure congestive (Cardiac disorders) | 1 | 4 | NA | NA
Cardiopulmonary failure (Cardiac disorders) | 1 | 0 | NA | NA
Coronary artery stenosis (Cardiac disorders) | 1 | 0 | NA | NA
Left ventricular dysfunction (Cardiac disorders) | 1 | 1 | NA | NA
Myocardial infarction (Cardiac disorders) | 3 | 4 | NA | NA
Palpitations (Cardiac disorders) | 2 | 0 | NA | NA
Pericardial effusion (Cardiac disorders) | 1 | 0 | NA | NA
Sinus node dysfunction (Cardiac disorders) | 0 | 1 | NA | NA
Tachycardia (Cardiac disorders) | 2 | 0 | NA | NA
Torsade de pointes (Cardiac disorders) | 0 | 1 | NA | NA
Sudden hearing loss (Ear and labyrinth disorders) | 0 | 1 | NA | NA
Adrenal insufficiency (Endocrine disorders) | 0 | 2 | NA | NA
Retinal detachment (Eye disorders) | 0 | 1 | NA | NA
Abdominal distension (Gastrointestinal disorders) | 0 | 2 | NA | NA
Abdominal hernia (Gastrointestinal disorders) | 1 | 0 | NA | NA
Abdominal pain (Gastrointestinal disorders) | 3 | 5 | NA | NA
Abdominal pain lower (Gastrointestinal disorders) | 0 | 1 | NA | NA
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | NA | NA
Anal fistula (Gastrointestinal disorders) | 1 | 0 | NA | NA
Anal ulcer haemorrhage (Gastrointestinal disorders) | 1 | 0 | NA | NA
Ascites (Gastrointestinal disorders) | 1 | 1 | NA | NA
Colitis (Gastrointestinal disorders) | 1 | 1 | NA | NA
Constipation (Gastrointestinal disorders) | 2 | 2 | NA | NA
Diarrhoea (Gastrointestinal disorders) | 5 | 10 | NA | NA
Duodenal ulcer (Gastrointestinal disorders) | 3 | 1 | NA | NA
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 0 | 2 | NA | NA
Enterocolitis (Gastrointestinal disorders) | 1 | 0 | NA | NA
Erosive oesophagitis (Gastrointestinal disorders) | 0 | 1 | NA | NA
Gastric fistula (Gastrointestinal disorders) | 1 | 0 | NA | NA
Gastric haemorrhage (Gastrointestinal disorders) | 0 | 1 | NA | NA
Gastritis (Gastrointestinal disorders) | 1 | 2 | NA | NA
Gastritis erosive (Gastrointestinal disorders) | 1 | 0 | NA | NA
Gastrointestinal disorder (Gastrointestinal disorders) | 1 | 0 | NA | NA
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 | 2 | NA | NA
Glossodynia (Gastrointestinal disorders) | 1 | 0 | NA | NA
Haematemesis (Gastrointestinal disorders) | 0 | 2 | NA | NA
Haematochezia (Gastrointestinal disorders) | 0 | 1 | NA | NA
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 | 1 | NA | NA
Ileus (Gastrointestinal disorders) | 3 | 0 | NA | NA
Inguinal hernia (Gastrointestinal disorders) | 2 | 1 | NA | NA
Intestinal obstruction (Gastrointestinal disorders) | 2 | 2 | NA | NA
Large intestine polyp (Gastrointestinal disorders) | 1 | 0 | NA | NA
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | NA | NA
Nausea (Gastrointestinal disorders) | 6 | 7 | NA | NA
Oesophagitis ulcerative (Gastrointestinal disorders) | 0 | 1 | NA | NA
Pancreatitis (Gastrointestinal disorders) | 5 | 2 | NA | NA
Pancreatitis acute (Gastrointestinal disorders) | 1 | 1 | NA | NA
Peptic ulcer (Gastrointestinal disorders) | 1 | 0 | NA | NA
Rectal haemorrhage (Gastrointestinal disorders) | 2 | 1 | NA | NA
Small intestinal haemorrhage (Gastrointestinal disorders) | 2 | 0 | NA | NA
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 2 | NA | NA
Stomatitis (Gastrointestinal disorders) | 0 | 1 | NA | NA
Swollen tongue (Gastrointestinal disorders) | 0 | 1 | NA | NA
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 | 1 | NA | NA
Vomiting (Gastrointestinal disorders) | 7 | 8 | NA | NA
Asthenia (General disorders) | 2 | 4 | NA | NA
Chest pain (General disorders) | 2 | 0 | NA | NA
Death (General disorders) | 1 | 0 | NA | NA
Disease progression (General disorders) | 1 | 1 | NA | NA
Fatigue (General disorders) | 3 | 12 | NA | NA
General physical health deterioration (General disorders) | 0 | 1 | NA | NA
Impaired healing (General disorders) | 1 | 0 | NA | NA
Malaise (General disorders) | 0 | 1 | NA | NA
Non-cardiac chest pain (General disorders) | 2 | 0 | NA | NA
Pain (General disorders) | 1 | 3 | NA | NA
Pneumatosis (General disorders) | 0 | 1 | NA | NA
Pyrexia (General disorders) | 5 | 13 | NA | NA
Sudden death (General disorders) | 0 | 1 | NA | NA
Cholecystitis (Hepatobiliary disorders) | 2 | 1 | NA | NA
Cholecystitis acute (Hepatobiliary disorders) | 1 | 2 | NA | NA
Cholelithiasis (Hepatobiliary disorders) | 2 | 1 | NA | NA
Drug-induced liver injury (Hepatobiliary disorders) | 1 | 2 | NA | NA
Gallbladder rupture (Hepatobiliary disorders) | 1 | 0 | NA | NA
Hepatic function abnormal (Hepatobiliary disorders) | 7 | 4 | NA | NA
Hepatitis (Hepatobiliary disorders) | 0 | 1 | NA | NA
Hepatotoxicity (Hepatobiliary disorders) | 8 | 0 | NA | NA
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 2 | NA | NA
Jaundice cholestatic (Hepatobiliary disorders) | 0 | 1 | NA | NA
Anaphylactic reaction (Immune system disorders) | 1 | 0 | NA | NA
Abscess (Infections and infestations) | 1 | 0 | NA | NA
Anal abscess (Infections and infestations) | 1 | 0 | NA | NA
Appendicitis (Infections and infestations) | 1 | 1 | NA | NA
Bacterial infection (Infections and infestations) | 0 | 1 | NA | NA
Bronchitis (Infections and infestations) | 1 | 0 | NA | NA
Cellulitis (Infections and infestations) | 1 | 1 | NA | NA
Complicated appendicitis (Infections and infestations) | 0 | 1 | NA | NA
Febrile infection (Infections and infestations) | 0 | 1 | NA | NA
Gastroenteritis (Infections and infestations) | 1 | 2 | NA | NA
H1N1 influenza (Infections and infestations) | 1 | 0 | NA | NA
Herpes zoster (Infections and infestations) | 0 | 1 | NA | NA
Infection (Infections and infestations) | 1 | 0 | NA | NA
Lower respiratory tract infection (Infections and infestations) | 0 | 2 | NA | NA
Otitis media (Infections and infestations) | 1 | 0 | NA | NA
Perinephric abscess (Infections and infestations) | 0 | 1 | NA | NA
Peritonitis (Infections and infestations) | 0 | 1 | NA | NA
Pneumocystis jirovecii pneumonia (Infections and infestations) | 1 | 0 | NA | NA
Pneumonia (Infections and infestations) | 7 | 6 | NA | NA
Pneumonia aspiration (Infections and infestations) | 0 | 1 | NA | NA
Pneumonia bacterial (Infections and infestations) | 0 | 1 | NA | NA
Pyelonephritis (Infections and infestations) | 1 | 0 | NA | NA
Pyelonephritis acute (Infections and infestations) | 0 | 1 | NA | NA
Renal abscess (Infections and infestations) | 0 | 1 | NA | NA
Retroperitoneal abscess (Infections and infestations) | 0 | 1 | NA | NA
Salmonella sepsis (Infections and infestations) | 0 | 1 | NA | NA
Sepsis (Infections and infestations) | 3 | 1 | NA | NA
Septic shock (Infections and infestations) | 1 | 0 | NA | NA
Urinary tract infection (Infections and infestations) | 3 | 1 | NA | NA
Wound infection (Infections and infestations) | 1 | 0 | NA | NA
Acetabulum fracture (Injury, poisoning and procedural complications) | 2 | 0 | NA | NA
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 1 | NA | NA
Brain herniation (Injury, poisoning and procedural complications) | 1 | 0 | NA | NA
Chemical poisoning (Injury, poisoning and procedural complications) | 0 | 1 | NA | NA
Contusion (Injury, poisoning and procedural complications) | 1 | 0 | NA | NA
Craniocerebral injury (Injury, poisoning and procedural complications) | 1 | 0 | NA | NA
Fall (Injury, poisoning and procedural complications) | 0 | 2 | NA | NA
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 | 0 | NA | NA
Femur fracture (Injury, poisoning and procedural complications) | 1 | 2 | NA | NA
Humerus fracture (Injury, poisoning and procedural complications) | 1 | 0 | NA | NA
Ilium fracture (Injury, poisoning and procedural complications) | 1 | 0 | NA | NA
Multiple fractures (Injury, poisoning and procedural complications) | 0 | 1 | NA | NA
Patella fracture (Injury, poisoning and procedural complications) | 0 | 1 | NA | NA
Tibia fracture (Injury, poisoning and procedural complications) | 1 | 0 | NA | NA
Alanine aminotransferase increased (Investigations) | 35 | 8 | NA | NA
Amylase increased (Investigations) | 0 | 1 | NA | NA
Aspartate aminotransferase increased (Investigations) | 17 | 2 | NA | NA
Blood alkaline phosphatase increased (Investigations) | 1 | 0 | NA | NA
Blood bilirubin increased (Investigations) | 2 | 2 | NA | NA
Blood calcium increased (Investigations) | 0 | 1 | NA | NA
Blood creatine increased (Investigations) | 1 | 0 | NA | NA
Blood creatine phosphokinase increased (Investigations) | 0 | 1 | NA | NA
Blood creatinine increased (Investigations) | 1 | 0 | NA | NA
Blood glucose decreased (Investigations) | 1 | 0 | NA | NA
Blood magnesium decreased (Investigations) | 0 | 1 | NA | NA
Blood potassium increased (Investigations) | 1 | 1 | NA | NA
Ejection fraction decreased (Investigations) | 1 | 1 | NA | NA
Electrocardiogram QT prolonged (Investigations) | 0 | 1 | NA | NA
Gamma-glutamyltransferase increased (Investigations) | 3 | 0 | NA | NA
Haemoglobin decreased (Investigations) | 1 | 0 | NA | NA
Hepatic enzyme increased (Investigations) | 6 | 1 | NA | NA
Lipase increased (Investigations) | 7 | 4 | NA | NA
Liver function test abnormal (Investigations) | 1 | 0 | NA | NA
Liver function test increased (Investigations) | 2 | 0 | NA | NA
Neutrophil count decreased (Investigations) | 2 | 0 | NA | NA
Platelet count decreased (Investigations) | 0 | 9 | NA | NA
Decreased appetite (Metabolism and nutrition disorders) | 2 | 2 | NA | NA
Dehydration (Metabolism and nutrition disorders) | 8 | 11 | NA | NA
Electrolyte imbalance (Metabolism and nutrition disorders) | 1 | 0 | NA | NA
Hyperamylasaemia (Metabolism and nutrition disorders) | 0 | 1 | NA | NA
Hypercalcaemia (Metabolism and nutrition disorders) | 5 | 1 | NA | NA
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1 | NA | NA
Hyperkalaemia (Metabolism and nutrition disorders) | 2 | 2 | NA | NA
Hyperlipasaemia (Metabolism and nutrition disorders) | 1 | 0 | NA | NA
Hyperuricaemia (Metabolism and nutrition disorders) | 1 | 2 | NA | NA
Hypocalcaemia (Metabolism and nutrition disorders) | 2 | 0 | NA | NA
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 1 | NA | NA
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0 | NA | NA
Hyponatraemia (Metabolism and nutrition disorders) | 4 | 7 | NA | NA
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 1 | NA | NA
Malnutrition (Metabolism and nutrition disorders) | 0 | 1 | NA | NA
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 0 | NA | NA
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 5 | NA | NA
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | NA | NA
Fistula (Musculoskeletal and connective tissue disorders) | 0 | 1 | NA | NA
Flank pain (Musculoskeletal and connective tissue disorders) | 2 | 1 | NA | NA
Groin pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | NA | NA
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | NA | NA
Intervertebral disc compression (Musculoskeletal and connective tissue disorders) | 0 | 1 | NA | NA
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 2 | NA | NA
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | NA | NA
Osteolysis (Musculoskeletal and connective tissue disorders) | 2 | 0 | NA | NA
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | NA | NA
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | NA | NA
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | NA | NA
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | NA | NA
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | NA | NA
Cholesteatoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | NA | NA
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | NA | NA
Endometrial cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | NA | NA
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | NA | NA
Haemangioblastoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | NA | NA
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | NA | NA
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | NA | NA
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | NA | NA
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2 | NA | NA
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | NA | NA
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | NA | NA
Metastasis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | NA | NA
Paraneoplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | NA | NA
Parathyroid tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | NA | NA
Renal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | NA | NA
Signet-ring cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | NA | NA
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | NA | NA
Tumour associated fever (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | NA | NA
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | NA | NA
Tumour rupture (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | NA | NA
Central nervous system haemorrhage (Nervous system disorders) | 1 | 1 | NA | NA
Cerebellar haemorrhage (Nervous system disorders) | 0 | 1 | NA | NA
Cerebral haemorrhage (Nervous system disorders) | 5 | 1 | NA | NA
Cerebral infarction (Nervous system disorders) | 0 | 2 | NA | NA
Cerebral ischaemia (Nervous system disorders) | 0 | 1 | NA | NA
Cerebral small vessel ischaemic disease (Nervous system disorders) | 0 | 1 | NA | NA
Cerebrovascular accident (Nervous system disorders) | 2 | 0 | NA | NA
Cerebrovascular insufficiency (Nervous system disorders) | 0 | 1 | NA | NA
Dizziness (Nervous system disorders) | 2 | 1 | NA | NA
Encephalopathy (Nervous system disorders) | 1 | 0 | NA | NA
Haemorrhage intracranial (Nervous system disorders) | 1 | 0 | NA | NA
Haemorrhagic cerebral infarction (Nervous system disorders) | 0 | 1 | NA | NA
Headache (Nervous system disorders) | 2 | 1 | NA | NA
Hemianaesthesia (Nervous system disorders) | 1 | 0 | NA | NA
Hypoaesthesia (Nervous system disorders) | 0 | 1 | NA | NA
Ischaemic stroke (Nervous system disorders) | 1 | 0 | NA | NA
Lethargy (Nervous system disorders) | 0 | 1 | NA | NA
Loss of consciousness (Nervous system disorders) | 0 | 1 | NA | NA
Metabolic encephalopathy (Nervous system disorders) | 1 | 0 | NA | NA
Motor dysfunction (Nervous system disorders) | 0 | 1 | NA | NA
Paraesthesia (Nervous system disorders) | 0 | 1 | NA | NA
Paraplegia (Nervous system disorders) | 1 | 0 | NA | NA
Presyncope (Nervous system disorders) | 0 | 1 | NA | NA
Seizure (Nervous system disorders) | 2 | 3 | NA | NA
Spinal cord compression (Nervous system disorders) | 4 | 3 | NA | NA
Subarachnoid haemorrhage (Nervous system disorders) | 0 | 1 | NA | NA
Syncope (Nervous system disorders) | 1 | 4 | NA | NA
Transient ischaemic attack (Nervous system disorders) | 3 | 1 | NA | NA
Tremor (Nervous system disorders) | 0 | 1 | NA | NA
Anxiety (Psychiatric disorders) | 0 | 1 | NA | NA
Confusional state (Psychiatric disorders) | 1 | 2 | NA | NA
Emotional distress (Psychiatric disorders) | 0 | 1 | NA | NA
Mental status changes (Psychiatric disorders) | 1 | 0 | NA | NA
Sleep disorder (Psychiatric disorders) | 0 | 1 | NA | NA
Acute kidney injury (Renal and urinary disorders) | 4 | 9 | NA | NA
Haematuria (Renal and urinary disorders) | 2 | 3 | NA | NA
Nephrotic syndrome (Renal and urinary disorders) | 0 | 1 | NA | NA
Proteinuria (Renal and urinary disorders) | 1 | 1 | NA | NA
Renal failure (Renal and urinary disorders) | 1 | 4 | NA | NA
Renal haemorrhage (Renal and urinary disorders) | 1 | 0 | NA | NA
Renal impairment (Renal and urinary disorders) | 0 | 1 | NA | NA
Ureteric obstruction (Renal and urinary disorders) | 1 | 0 | NA | NA
Urinary retention (Renal and urinary disorders) | 1 | 0 | NA | NA
Bartholin's cyst (Reproductive system and breast disorders) | 1 | 0 | NA | NA
Penile oedema (Reproductive system and breast disorders) | 1 | 0 | NA | NA
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | NA | NA
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | NA | NA
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | NA | NA
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5 | 8 | NA | NA
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 6 | NA | NA
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 3 | 2 | NA | NA
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | NA | NA
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | NA | NA
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | NA | NA
Laryngeal haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | NA | NA
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | NA | NA
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 11 | NA | NA
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | NA | NA
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | NA | NA
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | NA | NA
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | NA | NA
Pulmonary artery thrombosis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | NA | NA
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 8 | 7 | NA | NA
Pulmonary pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | NA | NA
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | NA | NA
Actinic keratosis (Skin and subcutaneous tissue disorders) | 0 | 1 | NA | NA
Angioedema (Skin and subcutaneous tissue disorders) | 1 | 0 | NA | NA
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1 | 0 | NA | NA
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 2 | 0 | NA | NA
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 | NA | NA
Aortic thrombosis (Vascular disorders) | 1 | 0 | NA | NA
Arterial rupture (Vascular disorders) | 0 | 1 | NA | NA
Deep vein thrombosis (Vascular disorders) | 2 | 0 | NA | NA
Dry gangrene (Vascular disorders) | 1 | 0 | NA | NA
Giant cell arteritis (Vascular disorders) | 0 | 1 | NA | NA
Haematoma (Vascular disorders) | 0 | 1 | NA | NA
Hypertension (Vascular disorders) | 7 | 6 | NA | NA
Hypertensive crisis (Vascular disorders) | 2 | 1 | NA | NA
Hypotension (Vascular disorders) | 1 | 1 | NA | NA
Orthostatic hypotension (Vascular disorders) | 0 | 1 | NA | NA
Thrombosis (Vascular disorders) | 1 | 1 | NA | NA
Vena cava thrombosis (Vascular disorders) | 1 | 1 | NA | NA
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Pazopanib 800 mg (N=554) | Sunitinib 50 mg (N=548) | Pazopanib 800 mg (Post-Treatment) (N=0) | Sunitinib 50 mg (Post-Treatment) (N=0)
Anaemia (Blood and lymphatic system disorders) | 36 | 99 | NA | NA
Leukopenia (Blood and lymphatic system disorders) | 51 | 100 | NA | NA
Neutropenia (Blood and lymphatic system disorders) | 60 | 147 | NA | NA
Thrombocytopenia (Blood and lymphatic system disorders) | 56 | 180 | NA | NA
Hyperthyroidism (Endocrine disorders) | 7 | 29 | NA | NA
Hypothyroidism (Endocrine disorders) | 71 | 138 | NA | NA
Eyelid oedema (Eye disorders) | 18 | 39 | NA | NA
Abdominal discomfort (Gastrointestinal disorders) | 24 | 33 | NA | NA
Abdominal distension (Gastrointestinal disorders) | 34 | 27 | NA | NA
Abdominal pain (Gastrointestinal disorders) | 72 | 74 | NA | NA
Abdominal pain upper (Gastrointestinal disorders) | 69 | 49 | NA | NA
Constipation (Gastrointestinal disorders) | 97 | 133 | NA | NA
Diarrhoea (Gastrointestinal disorders) | 349 | 312 | NA | NA
Dry mouth (Gastrointestinal disorders) | 26 | 29 | NA | NA
Dyspepsia (Gastrointestinal disorders) | 78 | 135 | NA | NA
Flatulence (Gastrointestinal disorders) | 32 | 15 | NA | NA
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 19 | 55 | NA | NA
Mouth ulceration (Gastrointestinal disorders) | 22 | 35 | NA | NA
Nausea (Gastrointestinal disorders) | 248 | 253 | NA | NA
Oral pain (Gastrointestinal disorders) | 12 | 28 | NA | NA
Stomatitis (Gastrointestinal disorders) | 78 | 154 | NA | NA
Vomiting (Gastrointestinal disorders) | 158 | 148 | NA | NA
Asthenia (General disorders) | 47 | 58 | NA | NA
Chills (General disorders) | 15 | 43 | NA | NA
Face oedema (General disorders) | 12 | 40 | NA | NA
Fatigue (General disorders) | 305 | 342 | NA | NA
Mucosal inflammation (General disorders) | 62 | 141 | NA | NA
Oedema (General disorders) | 15 | 37 | NA | NA
Oedema peripheral (General disorders) | 58 | 86 | NA | NA
Pyrexia (General disorders) | 47 | 77 | NA | NA
Nasopharyngitis (Infections and infestations) | 46 | 42 | NA | NA
Upper respiratory tract infection (Infections and infestations) | 30 | 34 | NA | NA
Urinary tract infection (Infections and infestations) | 23 | 29 | NA | NA
Alanine aminotransferase increased (Investigations) | 143 | 93 | NA | NA
Amylase increased (Investigations) | 39 | 24 | NA | NA
Aspartate aminotransferase increased (Investigations) | 128 | 96 | NA | NA
Blood alkaline phosphatase increased (Investigations) | 40 | 30 | NA | NA
Blood bilirubin increased (Investigations) | 51 | 35 | NA | NA
Blood creatinine increased (Investigations) | 52 | 85 | NA | NA
Blood lactate dehydrogenase increased (Investigations) | 40 | 60 | NA | NA
Blood thyroid stimulating hormone increased (Investigations) | 33 | 64 | NA | NA
Blood triglycerides increased (Investigations) | 21 | 35 | NA | NA
Haemoglobin decreased (Investigations) | 34 | 75 | NA | NA
Lipase increased (Investigations) | 43 | 32 | NA | NA
Neutrophil count decreased (Investigations) | 23 | 60 | NA | NA
Platelet count decreased (Investigations) | 36 | 97 | NA | NA
Weight decreased (Investigations) | 86 | 33 | NA | NA
White blood cell count decreased (Investigations) | 31 | 74 | NA | NA
Decreased appetite (Metabolism and nutrition disorders) | 207 | 203 | NA | NA
Hyperglycaemia (Metabolism and nutrition disorders) | 16 | 30 | NA | NA
Hyponatraemia (Metabolism and nutrition disorders) | 22 | 36 | NA | NA
Hypophosphataemia (Metabolism and nutrition disorders) | 21 | 32 | NA | NA
Arthralgia (Musculoskeletal and connective tissue disorders) | 98 | 82 | NA | NA
Back pain (Musculoskeletal and connective tissue disorders) | 91 | 89 | NA | NA
Flank pain (Musculoskeletal and connective tissue disorders) | 14 | 30 | NA | NA
Muscle spasms (Musculoskeletal and connective tissue disorders) | 38 | 23 | NA | NA
Myalgia (Musculoskeletal and connective tissue disorders) | 34 | 37 | NA | NA
Pain in extremity (Musculoskeletal and connective tissue disorders) | 70 | 93 | NA | NA
Dizziness (Nervous system disorders) | 71 | 82 | NA | NA
Dysgeusia (Nervous system disorders) | 49 | 58 | NA | NA
Headache (Nervous system disorders) | 124 | 122 | NA | NA
Taste disorder (Nervous system disorders) | 99 | 145 | NA | NA
Insomnia (Psychiatric disorders) | 58 | 61 | NA | NA
Haematuria (Renal and urinary disorders) | 24 | 28 | NA | NA
Proteinuria (Renal and urinary disorders) | 99 | 76 | NA | NA
Cough (Respiratory, thoracic and mediastinal disorders) | 86 | 105 | NA | NA
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 42 | 12 | NA | NA
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 79 | 92 | NA | NA
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 49 | 96 | NA | NA
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 39 | 54 | NA | NA
Alopecia (Skin and subcutaneous tissue disorders) | 77 | 45 | NA | NA
Dry skin (Skin and subcutaneous tissue disorders) | 44 | 47 | NA | NA
Hair colour changes (Skin and subcutaneous tissue disorders) | 168 | 54 | NA | NA
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 163 | 275 | NA | NA
Pruritus (Skin and subcutaneous tissue disorders) | 23 | 45 | NA | NA
Rash (Skin and subcutaneous tissue disorders) | 95 | 126 | NA | NA
Yellow skin (Skin and subcutaneous tissue disorders) | 4 | 93 | NA | NA
Hypertension (Vascular disorders) | 256 | 220 | NA | NA

LIMITATIONS AND CAVEATS:
This is a legacy GlaxoSmithKline (GSK) study and the primary CSR was completed by GSK prior to the study sponsorship handover. The full investigators lists and other appendices were not transferred over during the change in sponsorship from GSK to Novartis and therefore, the team could not confirm or quality control the investigator sites list.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.